CLINICAL TRIAL: NCT01572844
Title: Novel Drug Delivery of Sodium Thiosulfate for Calcinosis Associated With Adult and Juvenile Dermatomyositis
Brief Title: Topical Sodium Thiosulfate and Fractional Carbon Dioxide Laser in Treating Dermatomyositis Associated Calcinosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alison Ehrlich (Other)
Responsible Party: Sponsor-Investigator, Alison Ehrlich, Principal Investigator, George Washington University
Organization: George Washington University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 121131
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Calcinosis
Keywords: Dermatomyositis; Superficial calcinosis; Fractional carbon dioxide laser; Sodium thiosulfate
MeSH Terms: conditions — Calcinosis; Dermatomyositis | interventions — Lasers; sodium thiosulfate

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment lesion (Experimental): Lesion A, target lesion, 2cm x 2cm (+/- 1cm) treated with 1 pass Fractionated Carbon Dioxide (FCO2) Laser followed by application of 4 ml of 5% topical sodium thiosulfate solution (STS), 8 to 10 treatments over 6 months.
  Interventions: Device: Fractionated Carbon Dioxide (FCO2) Laser; Drug: Sodium thiosulfate
- No Treatment Lesion (No Intervention): Lesion B, similar area of calcinosis on the same patient, which did not receive treatment is evaluated.

INTERVENTIONS:
Device: Fractionated Carbon Dioxide (FCO2) Laser — At each treatment visit, a 2 X 2 cm (+/- 1 cm) area of the target calcinosis lesions will be treated with one pass of the Candela QuadraLase (TM) FCO2 laser. Patients will receive a total of 8-10 treatments over a 6 month period.
  Other Names: Candela QuadraLase (TM)
  Arms: Treatment lesion
Drug: Sodium thiosulfate — Following treatment with FCO2 laser, 4 ml of 5% Sodium Thiosulfate solution will be applied to the treatment site only. Subjects will receive a total of 8-10 treatments over a 6 month period.
  Arms: Treatment lesion

SUMMARY:
Dermatomyositis is an inflammatory muscle disorder that is often associated with many skin findings. One of the skin findings seen in up to 50% of individuals with juvenile dermatomyositis, an early onset form of this condition, and up to 20-30% of adult dermatomyositis patients who have not responded to treatment, is calcinosis, or deposits of calcium within the skin and muscle tissue. In addition to being cosmetically unappealing, involvement of deeper tissues with calcinosis may lead to contractures, or shortening of muscles, which may have a significant impact on functioning and quality of life. Unfortunately, there is no known effective treatment of dermatomyositis associated calcinosis. However, recent reports have shown that a medication called sodium thiosulfate has been effective in treating individuals with calciphylaxis, a condition where calcium is deposited within blood vessels, and with tumoral calcinosis, a genetic form of calcification, when receiving this medication by vein. In addition, recent advances in laser technology have led to the development of methods that may allow topical medications to penetrate deeper layers of the skin. The investigators have designed a pilot study to evaluate the use of topical sodium thiosulfate solution in treating superficial calcinosis in individuals with juvenile and adult dermatomyositis. The investigators will use laser to assist in the delivery of this medication to areas of calcinosis.

DETAILED DESCRIPTION:
Five individuals who meet the eligibility criteria will take part in this study. They will have a variety of assessments performed throughout the treatment period in order to evaluate both dermatomyositis and calcinosis severity and their potential response to fractional carbon dioxide and sodium thiosulfate treatment. A medical history will be taken and baseline assessments will be performed during the screening period. Serum creatinine kinase levels will be determined on this visit and repeated at the end of the study (week 20); these levels will be one measure of monitoring disease activity during the study. One calcinosis lesion will be treated, assessed, and followed. If a second calcinosis lesion is present, it will act as a control (not treated). Two weeks prior to the first treatment session, an optional (not required) skin biopsy of the target (treated) calcinosis lesion will be offered to the the first 3 patients ≥ 18 years of age to determine optimal fractional carbon dioxide laser settings that will be used for treatment. Area and durometer (a device that measures hardness) measurements and photographs of the calcinosis lesions will be performed at weeks 0,4,8,12,16,and 20. One x-ray of the control and one x-ray of the target calcinosis lesion will also be performed during the screening period and at week 20. Assessment of muscle strength, physical functioning, endurance, and range of motion, as well as myositis activity outside of the muscles will be performed during the screening period and at weeks 8 and 20. Myositis damage assessment will be performed at the screening period and at week 20. Questionnaires to assess physical functioning pertaining to activities of daily living and quality of life, as well as the quality of life related to skin disease and the calcinosis lesions will be completed during the screening period and at weeks 8 and 20. Treatment of the target calcinosis lesion with fractional carbon dioxide laser and topical sodium thiosulfate will occur on weeks 0,2,4,6,8,10,12,14,16,and 18. Each patient will receive a total of 8-10 treatments over a 6 month period. Assessments for any side effects from the treatment will be performed prior to each treatment session on weeks 0,2,4,6,8,10,12,14,16,18, and 20.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes and of all ethnicities who wish to participate in the study and who have signed a written informed consent form to participate.
* Subjects must be between the ages of 18-65 years.
* Subjects must have a diagnosis of adult or juvenile dermatomyositis.
* All patient must be on stable therapy for their condition. Overall disease activity must be considered mild or in remission.
* Patients must have a history of failing at least one therapy for calcinosis associated with dermatomyositis.
* Patients must have at least one localized area of superficial calcinosis with easily identifiable landmarks. Whenever possible, subjects will have a second localized area of superficial calcinosis that can serve as a control lesion for repeated assessment.
* The calcinosis lesion being treated and the control calcinosis lesion must be stable (not increasing in size) based on the patient's history.
* Patients must be able to attend all treatment sessions and assessment visits at our Washington, District of Columbia clinic over the 20 week period.

Exclusion Criteria:

* Unstable dermatomyositis, or moderate or severely active juvenile dermatomyositis.
* Serum creatine kinase greater than or equal to three times the upper limit of normal.
* Inability to make study visits or anticipated poor compliance.
* Active infections, including a history of recurrent superinfection or cellulitis at the sites of calcinosis (> 1 prior episode).
* Pregnant females or nursing mothers.
* Life threatening illness that would interfere with the patient's ability to complete the study.
* Known or suspected history of drug or alcohol abuse within the past 6 months.
* Participation in another clinical experimental therapeutic study within 30 days of screening visit.
* History of severe illness or any other condition that would make the patient unsuitable for the study.
* History of hepatitis B, hepatitis C, HIV, cancer-associated myositis, or an underlying malignancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Ehrlich, MD, Principal Investigator — George Washington University; Gary Simon, MD, Principal Investigator — George Washington University; James Katz, MD, Study Chair — George Washington University; Gulnara Mamayrova, MD, Study Chair — George Washington University; Laura Roosa, Study Chair — George Washington University; Andrea Morris, MD, Study Chair — George Washington University
Locations (1):
- The George Washington University Medical Faculty Associates Departments of Dermatology and Rheumatology, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants enrolled required 2 similar calcinosis lesions; one for the treatment arm and one for the no treatment arm.
Units Other Than Participants: lesion
Groups:
- Treatment Lesion: Lesion A, target lesion Fractionated Carbon Dioxide (FCO2) Laser: At each treatment visit, the target area (2cm x 2cm) (+/- 1cm) of the calcinosis lesions will be treated with one pass of the Candela QuadraLase (TM) FCO2 laser.
  Sodium thiosulfate: Following treatment with FCO2 laser, 4 ml of 5% Sodium Thiosulfate solution will be applied to the treatment site only.
  Subjects will receive a total of 8-10 treatments over a 6 month period.
- No Treatment Lesion: Lesion B, similar area of calcinosis on the same patient, which did not receive treatment, is evaluated.
Period: Overall Study
Arm/Group | Treatment Lesion | No Treatment Lesion
Started | 3; 3 lesion | 3; 3 lesion
Completed | 2; 2 lesion | 2; 2 lesion
Not Completed | 1; 1 lesion | 1; 1 lesion
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This Arm includes all participants who were enrolled in the study
Arm/Group | All Study Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Dermatomyositis-associated Calcinosis of a Single Lesion by Assessing Its Severity as Measured by a Difference in Physician Calcinosis Visual Analog Scales.
Description: Change in dermatomyositis-associated calcinosis of a single lesion by assessing its severity as measured by a difference in Physician Calcinosis Visual Analog Scales. The Visual Analog Scale range is from zero (0) to ten (10). Zero (0) being no evidence of disease activity and ten (10) being extremely active or severe disease activity. A negative percent change indicates improvement in the lesion.
Time Frame: Change from Visit 2 to Visit 12 (week 20)
Measure: Number; unit: percentage change
Units Other Than Participants: lesion
Arm/Group | Treatment Lesion | No Treatment Lesion
Number analyzed (Participants) | 2 | 2
Number analyzed (lesion) | 2 | 2
percentage change
  Subject 1 | -38.0 | 3.3
  Subject 2 | -53.1 | 2.0

2. Secondary Outcome: Change in Dermatomyositis-associated Calcinosis of a Single Lesion by Assessing Its Hardness as Measured by a Difference in Durometer (Rex Durometer Model 1600, Type OO) Measurements.
Description: Change in dermatomyositis-associated calcinosis of a single lesion by assessing its hardness as measured by a difference in durometer (Rex durometer Model 1600, Type OO) measurements. The range of a durometer is from 0 to 100. The higher the durometer reading, the harder the lesion. Improvement in the lesion hardness would result in a negative change over time.
Time Frame: Change from Baseline (Visit 1) at Final Assessment (Visit 12, week 20).
Population: 2 subjects were enrolled and each subject has 2 lesions that were followed through the study. Each subject has one area that was marked as treatment lesion and also has an area that was used as a control (no treatment lesion). Overall, there were 2 subjects, 2 treatment lesions and 2 no treatment lesions.
Measure: Number; unit: percentage of change
Units Other Than Participants: lesions
Groups:
- Treatment Lesion: Lesion A, target lesion Fractionated Carbon Dioxide (FCO2) Laser
Arm/Group | Treatment Lesion | No Treatment Lesion
Number analyzed (Participants) | 2 | 2
Number analyzed (lesions) | 2 | 2
percentage of change
  Subject 1 | -35.8 | -18.4
  Subject 2 | 7.4 | 23.8

3. Secondary Outcome: Change in Dermatomyositis-associated Calcinosis of a Single Lesion by Assessing Its Severity as Measured by a Difference in Patient Calcinosis Visual Analog Scales.
Description: Change in dermatomyositis-associated calcinosis of a single lesion by assessing its severity as measured by a difference in Patient Calcinosis Visual Analog Scales. The scale ranges from zero (0) to ten (10). Zero (0) being no evidence of disease activity and ten (10) being extremely active or severe disease activity. A negative change would indicate improvement in the disease activity. A positive change would indicate worsening of disease activity.
Time Frame: Change from Visit 2 to Visit 12 (week 20)
Measure: Number; unit: Percentage of change
Units Other Than Participants: lesions
Arm/Group | Treatment Lesion | No Treatment Lesion
Number analyzed (Participants) | 2 | 2
Number analyzed (lesions) | 2 | 2
Percentage of change
  Subject 1 | 104.7 | 136.5
  Subject 2 | 0 | 1.9

4. Secondary Outcome: Change in Size of Dermatomyositis-associated Calcinosis Area on Lesions as Measured by a Difference in Plain Film (X-ray) Studies.
Description: Change in dermatomyositis-associated calcinosis as measured by a difference in centimeters in plain film (x-ray) studies. X rays were compared between baseline and final assessment for any changes.
Time Frame: Change from Visit 2 to Visit 12 (week 20)
Population: No change was observed for any lesion.
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: lesion
Groups:
- Treatment Lesion: Lesion A, target lesion
- No Treatment Lesion: Lesion B, similar area of calcinosis on the same patient, which did not receive treatment
Arm/Group | Treatment Lesion | No Treatment Lesion
Number analyzed (Participants) | 2 | 2
Number analyzed (lesion) | 2 | 2
cm | 0 (0) | 0 (0)

5. Secondary Outcome: Change in Patient Functionality and/or Quality of Life.
Description: This will be assessed through the use of the Dermatology Life Quality Index (DLQI), Health Assessment Questionnaire (HAQ)/Childhood Health Assessment Questionnaire (CHAQ), Manual Muscle Testing (MMT8), and range of motion evaluations. DLQI index scores range from 0 to 30. The higher the score, the more quality of life is impaired.Change in scores from baseline to final assessment yielding a negative percent change indicate an improvement in DLQI. HAQ scales range from 0 to 3. The higher the score, the greater the disability. Change in scores from baseline to final assessment yielding a negative percent change indicate an improvement in the HAQ. MMT8 testing results in a score between 0 and 150. The higher the score, the more normal the function of the muscle. A positive percent change would indicate an improvement in MMT8 testing results.
Time Frame: Change from Visit 1 to Visit 12 (week 20)
Population: The arms/groups does not apply to this outcome measure. Lesions were not analyzed in these assessments. Overall Patient functionality and quality of life were evaluated via questionnaires, manual muscle testing, and range of motion evaluations. No changes in range of motion were noted for either subject.
Measure: Number; unit: percentage of change from baseline
Arm/Group | Treatment Lesion
Number analyzed (Participants) | 2
percentage of change from baseline
  DLQI : Subject 1 | -37.5
  DLQI : Subject 2 | 57.1
  HAQ : Subject 1 | -44.4
  HAQ : Subject 2 | 0
  MMT8 : Subject 1 | 3.4
  MMT8 : Subject 2 | -6.7

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the subjects' participation in the study, over a 6 month period.
Arm/Group | Treatment Lesion | No Treatment Lesion
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes